CLINICAL TRIAL: NCT01741649
Title: Clorhexidine Versus Povidone for the Prevention of Surgical Site Infection in Patients After Cesarean Section. Randomized, Controlled Trial.
Brief Title: Clorhexidine Versus Povidone for the Prevention of Surgical Site Infection After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHST2012-04
Record Dates: First submitted 2012-12-01; First posted 2012-12-05 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Surgical Wound Infection
Keywords: Surgical wound infection; Clorhexidine; Povidone
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clorhexidine (Experimental): Skin prior to the surgical incision will be cleaned for five minutes with Clorhexidine.
  Interventions: Procedure: Clorhexidine
- Povidone (Experimental): Skin prior to surgical incision will be cleaned for five minutes with a povidine solution.
  Interventions: Procedure: Povidone

INTERVENTIONS:
Procedure: Clorhexidine — Cleaning of the surgical site previous to the incision with a clorhexidine solution for five minutes.
  Arms: Clorhexidine
Procedure: Povidone — Cleaning of the surgical site previous to the incision with a povidone solution for five minutes.
  Arms: Povidone

SUMMARY:
Many solutions are used for cleaning the skin of a patient previous to a surgery. Although the efficacy of clorhexidine has been proved in other surgical procedures, there is only a retrospective study in cesarean section (they report no benefit of one solution over the other). The investigators would like to evaluate the difference in surgical site infection in patients after cesarean section comparing preparation of the skin with clorhexidine versus povidone.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 32 weeks
* Emergency cesarean section

Exclusion Criteria:

* Allergy to clorhexidine
* Allergy to povidone
* Evidence of infection in the surgical site
* Loss to follow up at 15 days
* Surgeries that due to the emergency of the case do not allow the five minutes of skin cleaning.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Surgical Site infection (SSI) | 3 days
  The patients will be evaluated for evidence of surgical site infection before leaving the hospital, three (3) days after surgery. The presence of fever, suppurative secretion through the wound or cutaneous changes compatible witn infection will be considered a surgical site infection (SSI). This outcome will be evaluated with a qualitative variable (presence of SSI). The patients will be classified in accordance as "With SSI" or "Without SSI".

SECONDARY OUTCOMES:
Hospitalization | 15 days
  The patients will be evaluated for evidence of surgical site infection 15 days post surgery. The need to admit the patient to the hospital for management of a surgical site infection will be classified with "Hospitalization - Yes/No".

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá, Panama